CLINICAL TRIAL: NCT05666063
Title: Comparison of Single Voiding Cycle and Two and Three Voiding Cycles in Ambulatory Urodynamic Studies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Bulut Varlı, Principal Investigator, Ankara University
Other Study IDs: AmbulatoryUDS-1
Record Dates: First submitted 2022-05-19; First posted 2022-12-27 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Urodynamics; Urinary Incontinence; Urogenital Disease, Female; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Incontinence; Female Urogenital Diseases; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients who underwent ambulatory urodynamic studies due to lower urinary tract symptoms
  Interventions: Diagnostic Test: Ambulatory Urodynamic Study

INTERVENTIONS:
Diagnostic Test: Ambulatory Urodynamic Study — Ambulatory urodynamic study is started after spontaneous diuresis of the patients. Ambulatory monitoring time is limited to each patient's own voiding cycle. The patient and a family member are instructed on the use of the event buttons on the patient module to flag incontinence, urgency, physical activity, and water drinking. With the use of catheters attached to microcomputers attached to their shoulders, patients are free to move around and engage in activities that may cause urinary incontinence. After voiding, the residual urine volume is first measured and then urethral and rectal catheters are placed. Monitoring is terminated when the patient feels that he cannot delay the urination sensation.Questionnaires that are routinely applied in our clinic will be applied in order to objectively evaluate the symptoms. Before urodynamics, urinary tract infection, whether symptomatic or not, must be routinely excluded with a complete urinalysis and urine culture.

SUMMARY:
Urodynamic studies are objective diagnostic methods recommended and used in the evaluation and diagnosis of urinary incontinence, which is a very common problem that can significantly affect women's health and quality of life, cause social and economic losses. With these examinations, objective observation of bladder functions, repetition and classification of patients' symptoms, and identification of the underlying pathological cause, if possible, are provided in the evaluation of lower urinary system dysfunctions; In this way, the diagnosis is made, the choice of treatment is affected, the results of the treatment can be predicted and appropriate counseling can be given to the patients. Although conventional urodynamics is currently accepted as the gold standard test in the investigation of lower urinary tract symptoms, non-physiological retrograde bladder filling may adversely affect the test results and patients have to be under observation on the examination table while being examined with the conventional urodynamic method. Conventional method may not be effective enough in revealing the etiopathogenesis of lower urinary system symptoms, because they cannot perform activities where lower urinary system symptoms occur. Although many studies have shown that the diagnostic value of ambulatory urodynamics (AU) is higher in urogynecology clinical practice, it was not found suitable for routine investigation due to its longer duration, time-consuming and cost-effectiveness. For this reason, its routine use has been limited in international guidelines for AU in cases where conventional urodynamics is insufficient in the diagnosis, by indicating its application. In the AU method, all physiopathological changes in the lower urinary system can be observed synchronously, since the bladder filling is orthograde, not retrograde, that is, the lower urinary system is examined while the physiological urine is filled, not liquid, and the patients can perform the activities they want, and the symptoms that occur during these activities can be recorded by the patient. Despite the advantages of performing it under these conditions, it takes a long time to be evaluated with 2-4 voiding cycles and is used as a second step in cases that cannot be diagnosed by conventional urodynamics. In the previous studies performed by us, it was seen that the results of the ambulatory urodynamic examination performed with a single voiding cycle were similar to the studies in the literature using multiple voiding cycles. However, at the moment, there is no study in the literature that determines the optimal duration of this test. For these reasons, this study aimed to compare the effectiveness of the test at the end of a single voiding cycle with that at the end of multiple (2 to 4) voiding cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. No suspicion of pregnancy
3. Adequate mental functions
4. Cases of stress urinary incontinence not confirmed by cough testing
5. Having inconsistent examination results
6. Significant urge, urge incontinence and/or overactive bladder complaints
7. Cases with mixed-type urinary incontinence with a predominant complaint of urgency
8. Those with a history of pelvic organ prolapse repair surgery
9. Those with a history of anti-incontinence surgery

Exclusion Criteria:

1. Presence of active urinary tract infection
2. Patients to be treated conservatively
3. Presence of urinary retention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological female patients
Study Population: Patients who applied to Ankara University Faculty of Medicine, Department of Obstetrics and Gynecology with complicated urinary system symptoms detected by anamnesis and physical examination will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy and feasibility | 2 year
  Determination of efficacy of single voiding cycle ambulatory urodynamics in diagnosis of lower urinary tract disorders by comparing number of incontinence and urgency episodes during the urodynamic study period

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No